CLINICAL TRIAL: NCT03444272
Title: Effect of Direct-acting Antiviral Drugs on Erectile Function Among Hepatitis c Patients
Brief Title: Effect of Direct-acting Antiviral Drugs on Erectile Function
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Collaborators: Benha University (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, PhDTropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCV TREATMENT
Record Dates: First submitted 2018-02-19; First posted 2018-02-23 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hepatitis C Treatment (Experimental): HCV Treatment (Sofosbuvir and Daklatasuvir)
  Interventions: Drug: Sofosbuvir and Daklatasuvir
- Supportive treatment (No Intervention): supportive liver therapy

INTERVENTIONS:
Drug: Sofosbuvir and Daklatasuvir — HCV Treatment (Sofosbuvir and Daklatasuvir)
  Other Names: Sofaldy, mpiviropack, daklanork
  Arms: Hepatitis C Treatment

SUMMARY:
Effect of direct-acting antiviral drugs on erectile function

DETAILED DESCRIPTION:
Effect of direct-acting antiviral drugs on erectile function in HCV patients

ELIGIBILITY:
Inclusion Criteria:

* HCV infected patients
* Male

Exclusion Criteria:

* HCC
* Age below 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males
Enrollment: 105 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with improved erectile functions | 6 months
  Number of patients with improved erectile functions

CONTACTS AND LOCATIONS:
Overall Officials: Sherief Abd-Elsalam, MD, Study Chair — Tanta University; Mohamed Alhefnawy, MD, Principal Investigator — Tanta University Faculty of medicine; Khaled Almekaty, MD, Principal Investigator — Tanta University
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided